CLINICAL TRIAL: NCT05578209
Title: Therapeutic Impacts of Theta Burst Stimulation Over Bilateral Posterior Superior Temporal Sulcus in Autism Spectrum Disorder: a Comprehensive Study Integrating Clinical Symptoms, Neuropsychological Function and MRI
Brief Title: Therapeutic Impacts of Theta Burst Stimulation Over Bilateral Posterior Superior Temporal Sulcus in Autism Spectrum Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202102232A0
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): Participants received the intervention of iTBS (The total pulse of every session is 1200 pulses) over bilateral posterior superior temporal sulcus for 4 weeks (5 days/week).
  *iTBS = intermittent theta burst stimulation
  Interventions: Device: intermittent theta burst stimulation
- Sham (Sham Comparator): Participants received the sham intervention of iTBS (sham-coil) over bilateral posterior superior temporal sulcus for 4 weeks (5 days/week).
  Interventions: Device: intermittent theta burst stimulation

INTERVENTIONS:
Device: intermittent theta burst stimulation — stimulatory protocol

SUMMARY:
The investigator would like to investigate the impact of intermittent theta burst stimulation over bilateral posterior superior temporal sulcus in autism spectrum disorder

ELIGIBILITY:
Inclusion Criteria:

* Autism spectrum disorder, confirmed by Autism Diagnostic Observation Schedule II (CSS≧6)
* No change in psychiatric drugs within one month

Exclusion Criteria:

* Previous or current severe neurological disorder such as epilepsy, visual or hearing impairment
* Previous or current severe systemic disease such as cardiovascular disease, diabetes or infection
* Previous or current severe brain injury
* Implementation of metal materials such as pacemaker or medication pump
* Previous or current severe psychiatric disorders such as schizophrenia, bipolar disorder or substance abuse
* Pregnancy
* Individuals with a significant brain abnormality such as intracranial space occupied lesions
* History of brain surgery or nervous system infection, such as meningitis and encephalitis
* Previous febrile seizures
* Concurrent use of medications which increased the risk of seizure attack.
* Participate another clinical trial within one month.
* Unable to complete MRI scan (claustrophobia)
* Skin trauma on application site
* Individuals with a large ischemic scar
* Individuals suffering from multiple sclerosis
* Individuals suffering from sleep deprivation during rTMS procedures
* Individuals with a heavy consumption of alcohol
* Individuals with a migraine headache from increased intracranial pressure

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of total scores of Social Responsiveness Scale | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.
Changes of total scores of Repetitive Behavior Scale-Revised | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  Repetitive Behavior Scale-Revised is a questionnaire that focuses on repetitive behavior. The score ranges from 0-129. The lower scores stand for lower repetitive behavior.

SECONDARY OUTCOMES:
Changes of total scores of Aberrant Behavior Checklist | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  ABC is a parents' report questionnaire for aberrant behavior. The lower scores stand for less aberrant behavior.
Changes of total scores of Emotional Dysregulation Inventory | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  Emotional Dysregulation Inventory is a parents' report questionnaire for emotional dysregulation. The score ranges from 0-120. The lower scores stand for better emotional regulation.
Changes of total scores of Child Behavior Checklist | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  CBCL is a parents' report questionnaire for behavioral and emotional problems. The lower scores stand for better behavioral and emotional regulation.
Changes of total scores of Adaptive Behavior Assessment System | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  Adaptive Behavior Assessment System is a parents' report questionnaire for adaptive behavior. The score ranges from 9-171. The higher scores stand for better adaptive behavior.
Changes in accuracy of Frith-Happe animation | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition.
Changes in accuracy of Eyes task | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills.
Changes in accuracy of Wisconsin Card Sorting Test | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  An advanced test for cognitive flexibility. 128 questions in total, the more correct questions stand for better cognitive flexibility.
Changes of total scores of Behavior Rating Inventory of Executive Function | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  An advanced test for cognitive flexibility. 128 questions in total, the more correct questions stand for better cognitive flexibility.
Raven's Progressive Matrices | baseline; post TBS (4 weeks after baseline); One month follow up (8 weeks after baseline); Two months follow up (12 weeks after baseline)
  An advanced test for for executive function. 60 questions in total, the more correct questions stand for better executive function.
MRI T1 | baseline; post TBS (4 weeks after baseline)
  Brain structural volumes (cm²)
functional MRI (resting-state/biological motion task) - BOLD signal | baseline; post TBS (4 weeks after baseline)
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.
Diffusion Tensor Imaging (DTI) - FA | baseline; post TBS (4 weeks after baseline)
  Fractional anisotropy (FA) is a measurement used in DTI, which reflects the movement of water molecules. FA ranges from 0 to 1, the higher FA value may represent more intact axons.
Electroencephalography | baseline; post TBS (4 weeks after baseline)
  Resting state EEG (alpha power / frontal gamma power)

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan